CLINICAL TRIAL: NCT04197440
Title: Characterization of Bovine Adrenal Medulla (BAM8-22) as a New Surrogate Model of Non-histaminergic Itch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Giulia Erica Aliotta, PhD fellow, Aalborg University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20190062
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — bovine adrenal medulla 8-22

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bam8-22 (Experimental)
  Interventions: Drug: BAM8-22 2mg/ml; Drug: BAM8-22 1mg/ml; Drug: BAM8-22 0.5 mg/ml; Drug: Placebo
- SPT pricks (Experimental)
  Interventions: Drug: BAM8-22 with 1 SPT; Drug: BAM8-22 with 5 SPT; Drug: BAM8-22 with 25 SPT; Drug: BAM8-22 with inactivate cowhage spicules

INTERVENTIONS:
Drug: BAM8-22 2mg/ml — 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Arms: Bam8-22
Drug: BAM8-22 1mg/ml — 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Arms: Bam8-22
Drug: BAM8-22 0.5 mg/ml — 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Arms: Bam8-22
Drug: Placebo — 20 µl of water will be applied to a previously determined area on the volar forearm followed by a prick through the drop
  Arms: Bam8-22
Drug: BAM8-22 with 1 SPT — 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by 1 prick through the drop
  Arms: SPT pricks
Drug: BAM8-22 with 5 SPT — 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by 5 prick through the drop
  Arms: SPT pricks
Drug: BAM8-22 with 25 SPT — 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm followed by 25 prick through the drop
  Arms: SPT pricks
Drug: BAM8-22 with inactivate cowhage spicules — 20 µl of BAM8-22 will be applied to a previously determined area on the volar forearm using inactivate cowhage spicules
  Arms: SPT pricks

SUMMARY:
With this experiment, the experimenter wish to create a new model of itch based on the substance BAM8-22 (Bovine Adrenal Medulla), which is found naturally in the human body and which has proved to evoke itch.

DETAILED DESCRIPTION:
With this experiment, the experimenter wish to create a new model of itch based on the substance BAM8-22 (Bovine Adrenal Medulla), which is found naturally in the human body and which has proved to evoke itch.To explore and validate the dose-response features of a of this new itch model based on BAM8-22.

The experimenter will also characterize the sensory quality and temporary aspects of BAM8-22 skin prick test (SPT) in comparison to the inactivated-cowhage delivery system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current history of neurological, dermatological, immunological musculoskeletal, cardiac disorder or mental illnesses that may affect the results (e.g. neuropathy, muscular pain in the upper extremities, etc.)
* Moles, wounds, scars or tattoos in the area to be treated or tested
* Lack of ability to cooperate •
* Current use of medications that may affect the trial such as antihistamines and pain killers.
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these - Acute or chronic pain •
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
superficial blood perfusion | change from baseline, up to 10 minutes after the first session
  is measured by a speckle contrast imager (FLPI, Moor Instruments, England)
Warm Detection Threshold, and Heat Pain threshold | change from baseline, up to 10 minutes after the first session
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Cold Detection Threshold and Cold Pain threshold | change from baseline, up to 10 minutes after the first session
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Pain supra-threshold heat Stimuli | change from baseline, up to 10 minutes after the first session
  the tests for thermal sensation will all be performed using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device
Alloknesis | change from baseline, up to 10 minutes after the first session
  is measured by using a mildy pruritic, non-painful von Frey filaments of a predetermined intensity (generally 5-30 milliNewton of force)
mechanical pain threshold and sensitivity | change from baseline, up to 10 minutes after the first session
  is performed using a pin-prick set (Aalborg University). The set consists of 8 needles each having a diameter of 0,6 mm and different force applications
itch rating | change from baseline, up to 10 minutes after the first session
  the subject will rate the itch for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no itch" and 100 indicates "worst imaginable itch"

SECONDARY OUTCOMES:
pain rating | change from baseline, up to 10 minutes after the first session
  the subject will rate the pain for 10 minutes by using a visual analog scale (VAS) on a tablet. this scale goes from 0 to 100. 0 indicates "no pain" and 100 indicates "worst imaginable pain"

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark